CLINICAL TRIAL: NCT00002902
Title: PHASE I TRIAL OF IRINOTECAN AND TOMUDEX IN COMBINATION ON AN EVERY THREE WEEK SCHEDULE
Brief Title: Irinotecan Plus ICI D1694 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065242; UPCC-T96-0063; JMC-T96-0063; NCI-T96-0063O
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2002-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan; raltitrexed

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: raltitrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of irinotecan plus ICI D1694 in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of ICI D1694 (TDX) when given with irinotecan (CPT-11) every 3 weeks in patients with advanced solid malignancies. II. Describe the pharmacokinetics of TDX and CPT-11 when given in combination. III. Investigate the relationship between topoisomerase I expression in peripheral mononuclear cells and myelosuppression and/or gastrointestinal toxicity. IV. Investigate the effect of CPT-11 on thymidylate synthase expression in tumor.

OUTLINE: This is a dose-escalating study to determine the maximum tolerated dose (MTD) of ICI D1694 (TDX) given in combination with irinotecan. Irinotecan is given intravenously on day 1 and ICI D1694 intravenously on day 2. Treatment is repeated every 3 weeks until disease progression or unacceptable toxicity intervenes. Cohorts of 3-6 patients receive escalated doses of TDX until the MTD is defined; an additional 10-12 patients will be entered at the MTD to confirm this as a recommended phase II dose.

PROJECTED ACCRUAL: 30-35 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumor for which no effective therapy exists Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Hematopoietic: WBC at least 3,000 AGC at least 1,500 Platelets at least 100,000 Hepatic: Bilirubin no greater than 1.5 mg/dL AST/ALT no greater than 5 times normal Renal: Creatinine no greater than 1.5 mg/dL Metabolic: Glucose no greater than 200 mg/dL Electrolytes within 10% normal Other: No active infection that contraindicates entry No significant medical problem that contraindicates entry Effective contraception required of fertile patients Able and willing to participate in pharmacokinetic sampling

PRIOR CONCURRENT THERAPY: At least 3 weeks since chemotherapy (6 weeks since mitomycin or nitrosoureas) and recovered At least 3 weeks since radiotherapy and recovered

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. O'Dwyer, MD, BCh, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania, United States